CLINICAL TRIAL: NCT06199999
Title: A Randomized Controlled Trial Comparing the Effect of Erector Spinae Plane Blocks Versus High Volume Local Infiltration Analgesia on Pain, Inflammation and Cognitive Outcomes Following Thoraco-Lumbar Fusion Surgery
Brief Title: Erector Spinae Plane Block vs Local Infiltration Following Fusion Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rashmi Mueller (Other)
Responsible Party: Sponsor-Investigator, Rashmi Mueller, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202201643
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Delirium; Pain, Postoperative; Degenerative Disc Disease
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative; Intervertebral Disc Degeneration | interventions — Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group GA: General anesthesia only (No Intervention): This group receives general anesthesia only and surgical procedure will follow standard conditions.
- Group ESP: Erector Spinae Block (Active Comparator): This group receives general anesthesia with regional pain block (Erector Spinae Block) prior to incision.
  Interventions: Procedure: Erector Spinae Block
- Group LIA: Local Infiltration (Active Comparator): This group receives general anesthesia and surgical procedure will take place as planned. Prior to being awakened, the area of procedure will be infiltrated.
  Interventions: Procedure: Local infiltration with local anesthetic

INTERVENTIONS:
Procedure: Erector Spinae Block — General anesthesia with Erector Spinae Plane Block
  Arms: Group ESP: Erector Spinae Block
Procedure: Local infiltration with local anesthetic — General anesthesia with local infiltration of local anesthetic:
  Arms: Group LIA: Local Infiltration

SUMMARY:
The proposed intervention will examine two alternative methods for postoperative pain control. Two treatment arms of this study will include subjects who receive an erector spinae block (ESP) after induction of anesthesia but prior to the start of surgery and subjects who will receive a high volume of local anesthetic infiltration at the end of the procedure before emergence from anesthesia. The control group of subjects will undergo spinal surgery with general anesthesia but without any regional anesthesia. Outcome measurements include evaluation of serum inflammatory markers, pain scores, opioid usage and standardized evidence-based assessment methodologies.

DETAILED DESCRIPTION:
Treatment arms include:

* Group ESP (Erector Spinae Plane). This group receives general anesthesia with ESP (Erector Spinae Block) regional pain block prior to incision.
* Group LIA (Local Infiltration Anesthesia). This group receives general anesthesia and surgical procedure will take place as planned. Prior to being awakened, the area of procedure will be infiltrated using local anesthetic (LIA).
* Group GA. This group receives general anesthesia (GA) only and surgical procedure will follow standard conditions.

Pre-procedure activities for all groups will include survey evaluations. If the surveys demonstrate pre-procedure cognitive deficits, the subject's participation will cease.

All subjects who do not display deficits will complete baseline evaluations that include social history, pain medication history and rate their pain (scored from 1 to 10). The subjects will be randomized to a treatment group. Once the subject is asleep and prior to incision, laboratory blood tests will be drawn and again approximately 24 hours after the subject is received into the recovery unit. Following their surgical procedure, pain control for all subjects will be at the discretion of their primary care team. However, as part of the study, the amount of opioid medications required to control their pain and their pain rating score for the first 72 hours post surgery will be collected from the subject's medical record unless discharged from the hospital before this cutoff time. On post-operative days when subject remains in the hospital facility, repeat survey evaluations will be carried out and during the first 7 days of the subject's hospital stay and unanticipated event will be recorded from the subject's medical record.

ELIGIBILITY:
Inclusion Criteria for all groups:

1. Age: Greater than 18 years but less than 80
2. Surgical procedure: 1 to 2 level thoraco-lumbar fusion between T8 and S2; non-emergent surgery
3. Opioid naive (less than 6 oxycodone/day or 30 mg oxycodone equivalent)
4. No contraindication to local anesthetics or regional procedures.

Exclusion Criteria for all groups:

1. Emergency surgery
2. Allergy to study medications
3. BMI less than 20 or greater than 50
4. Major liver or kidney dysfunction or other pre-existing major organ dysfunction
5. Revision surgery
6. Opioid tolerant (60 mg morphine equivalents/day for 1 week) or narcotic dependence (opioid intake morphine equivalent greater than10 mg/day for more than 3 months)
7. Other sources of chronic pain (e.g. fibromyalgia)
8. Patients with associated significant central nervous system (CNS) or respiratory disease (home oxygen use)
9. Pre-operative neurological deficits
10. Co-existing hematological disorders or deranged coagulation parameters
11. Significant psychiatric illnesses that impedes the subject's ability to provide informed consent
12. Language barrier
13. Vulnerable population (e.g. prisoners)
14. Pregnant females
15. History of recent myocardial infarction
16. History of recent cardiac stent procedure (within 3 months)
17. Cardiac ejection fraction < 30%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of Quality of Recovery (QoR-15) Scores Between Treatment Groups | Change from pre-operation score to 1 day after surgery date
  The Quality of Recovery-15 (QoR-15) is a patient reported assessment aimed to validate the patients recovery following surgical intervention. The subject is asked to provide a quantitative number to a series of questions. The answers are rated on a scale from 0 to 10, where 0 = none of the time and 10 = all of the time. The scores for all of the questions are summed and comparison between the treatment groups will be assessed.
Quantitate the Change in Delirium Symptoms; Pre- to post-operative day 1 | Change from pre-operation score to 1 day after surgery date
  Potential new onset of delirium following surgical procedure will be assessed using the standardized 3D CAM ASSESSMENT (3-Minute Diagnostic Interview for the Confusion Assessment Method (CAM)). The subject is asked a series of questions and their responses are recorded. This structured mental status assessment is designed to detect the presence or absence of delirium. "The CAM algorithm is considered positive if the following features are present: Feature 1) Acute onset or fluctuating course and Feature 2) Inattention and either Feature 3) Disorganized thinking or Feature 4) Altered level of consciousness."
  Comparison between the treatment groups will be assessed and the presence of post-operative delirium reported.
  Reference: Marcantonio et al., (PMID: 25329203) and training manual.

SECONDARY OUTCOMES:
Quantitate the Change in Delirium Symptoms; Pre- to post-operative day 3 | Change from pre-operation score to 3 days after surgery date
  Potential new onset of delirium following surgical procedure will be assessed using the standardized 3D CAM ASSESSMENT (3-Minute Diagnostic Interview for the Confusion Assessment Method (CAM)). The subject is asked a series of questions and their responses are recorded. This structured mental status assessment is designed to detect the presence or absence of delirium. "The CAM algorithm is considered positive if the following features are present: Feature 1) Acute onset or fluctuating course and Feature 2) Inattention and either Feature 3) Disorganized thinking or Feature 4) Altered level of consciousness."
  Comparison between the treatment groups will be assessed and the presence of post-operative delirium reported.
  Reference: Marcantonio et al., (PMID: 25329203) and training manual.

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Mueller, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Health Care Medical Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be shared with researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual participant data (IPD) will be available for sharing immediately after publication and ending 5 years following article publication.
Access Criteria: Individual participant data (IPD) will be accessible to researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal.

REFERENCES:
- [Background] Brown CH 4th, LaFlam A, Max L, Wyrobek J, Neufeld KJ, Kebaish KM, Cohen DB, Walston JD, Hogue CW, Riley LH. Delirium After Spine Surgery in Older Adults: Incidence, Risk Factors, and Outcomes. J Am Geriatr Soc. 2016 Oct;64(10):2101-2108. doi: 10.1111/jgs.14434. Epub 2016 Oct 3. PMID 27696373
- [Background] Dunne SS, Coffey JC, Konje S, Gasior S, Clancy CC, Gulati G, Meagher D, Dunne CP. Biomarkers in delirium: A systematic review. J Psychosom Res. 2021 Aug;147:110530. doi: 10.1016/j.jpsychores.2021.110530. Epub 2021 Jun 1. PMID 34098376
- [Background] Ehrlich GE. Low back pain. Bull World Health Organ. 2003;81(9):671-6. Epub 2003 Nov 14. PMID 14710509
- [Background] Etzioni DA, Liu JH, O'Connell JB, Maggard MA, Ko CY. Elderly patients in surgical workloads: a population-based analysis. Am Surg. 2003 Nov;69(11):961-5. PMID 14627256
- [Background] Fineberg SJ, Nandyala SV, Marquez-Lara A, Oglesby M, Patel AA, Singh K. Incidence and risk factors for postoperative delirium after lumbar spine surgery. Spine (Phila Pa 1976). 2013 Sep 15;38(20):1790-6. doi: 10.1097/BRS.0b013e3182a0d507. PMID 23797502
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Huang X, Wang J, Zhang J, Kang Y, Sandeep B, Yang J. Ultrasound-guided erector spinae plane block improves analgesia after laparoscopic hepatectomy: a randomised controlled trial. Br J Anaesth. 2022 Sep;129(3):445-453. doi: 10.1016/j.bja.2022.05.013. Epub 2022 Jul 6. PMID 35803754
- [Background] Hughey AB, Lesniak MS, Ansari SA, Roth S. What will anesthesiologists be anesthetizing? Trends in neurosurgical procedure usage. Anesth Analg. 2010 Jun 1;110(6):1686-97. doi: 10.1213/ANE.0b013e3181cbd9cc. Epub 2010 Feb 8. PMID 20142356
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Kendall MC, Alves L, Traill LL, De Oliveira GS. The effect of ultrasound-guided erector spinae plane block on postsurgical pain: a meta-analysis of randomized controlled trials. BMC Anesthesiol. 2020 May 1;20(1):99. doi: 10.1186/s12871-020-01016-8. PMID 32357842
- [Background] Kumar CD, Dietz N, Sharma M, Cruz A, Counts CE, Wang D, Ugiliweneza B, Boakye M, Drazin D. Spine Surgery in the Octogenarian Population: A Comparison of Demographics, Surgical Approach, and Healthcare Utilization With the PearlDiver Database. Cureus. 2021 Apr 19;13(4):e14561. doi: 10.7759/cureus.14561. PMID 34026377
- [Background] Lang SAJ, Bohn T, Barleben L, Pumberger M, Roll S, Buttner-Janz K. Advanced meta-analyses comparing the three surgical techniques total disc replacement, anterior stand-alone fusion and circumferential fusion regarding pain, function and complications up to 3 years to treat lumbar degenerative disc disease. Eur Spine J. 2021 Dec;30(12):3688-3701. doi: 10.1007/s00586-021-06784-6. Epub 2021 Apr 10. PMID 33837832
- [Background] Leslie K, Troedel S, Irwin K, Pearce F, Ugoni A, Gillies R, Pemberton E, Dharmage S. Quality of recovery from anesthesia in neurosurgical patients. Anesthesiology. 2003 Nov;99(5):1158-65. doi: 10.1097/00000542-200311000-00024. PMID 14576554
- [Background] Li K, Ji C, Luo D, Feng H, Yang K, Xu H. Wound infiltration with ropivacaine as an adjuvant to patient controlled analgesia for transforaminal lumbar interbody fusion: a retrospective study. BMC Anesthesiol. 2020 Nov 18;20(1):288. doi: 10.1186/s12871-020-01205-5. PMID 33208089
- [Background] Ma J, Bi Y, Zhang Y, Zhu Y, Wu Y, Ye Y, Wang J, Zhang T, Liu B. Erector spinae plane block for postoperative analgesia in spine surgery: a systematic review and meta-analysis. Eur Spine J. 2021 Nov;30(11):3137-3149. doi: 10.1007/s00586-021-06853-w. Epub 2021 May 13. PMID 33983515
- [Background] Mukherjee I. Invited commentary on "Effects of erector spinae plane block on postoperative pain and side-effects in adult patients underwent surgery: A systematic review and meta-analysis of randomized controlled trials". Int J Surg. 2020 Aug;80:35. doi: 10.1016/j.ijsu.2020.06.028. Epub 2020 Jun 22. No abstract available. PMID 32585193
- [Background] Nazemi AK, Gowd AK, Carmouche JJ, Kates SL, Albert TJ, Behrend CJ. Prevention and Management of Postoperative Delirium in Elderly Patients Following Elective Spinal Surgery. Clin Spine Surg. 2017 Apr;30(3):112-119. doi: 10.1097/BSD.0000000000000467. PMID 28141603
- [Background] Perera AP, Chari A, Kostusiak M, Khan AA, Luoma AM, Casey ATH. Intramuscular Local Anesthetic Infiltration at Closure for Postoperative Analgesia in Lumbar Spine Surgery: A Systematic Review and Meta-Analysis. Spine (Phila Pa 1976). 2017 Jul 15;42(14):1088-1095. doi: 10.1097/BRS.0000000000001443. PMID 28426530
- [Background] Rizk P, Morris W, Oladeji P, Huo M. Review of Postoperative Delirium in Geriatric Patients Undergoing Hip Surgery. Geriatr Orthop Surg Rehabil. 2016 Jun;7(2):100-5. doi: 10.1177/2151458516641162. Epub 2016 Apr 18. PMID 27239384
- [Background] Rizkalla JM, Holderread B, Awad M, Botros A, Syed IY. The erector spinae plane block for analgesia after lumbar spine surgery: A systematic review. J Orthop. 2021 Feb 18;24:145-150. doi: 10.1016/j.jor.2021.02.006. eCollection 2021 Mar-Apr. PMID 33716419
- [Background] Rudolph JL, Inouye SK, Jones RN, Yang FM, Fong TG, Levkoff SE, Marcantonio ER. Delirium: an independent predictor of functional decline after cardiac surgery. J Am Geriatr Soc. 2010 Apr;58(4):643-9. doi: 10.1111/j.1532-5415.2010.02762.x. Epub 2010 Mar 22. PMID 20345866
- [Background] Saadawi M, Layera S, Aliste J, Bravo D, Leurcharusmee P, Tran Q. Erector spinae plane block: A narrative review with systematic analysis of the evidence pertaining to clinical indications and alternative truncal blocks. J Clin Anesth. 2021 Feb;68:110063. doi: 10.1016/j.jclinane.2020.110063. Epub 2020 Oct 5. PMID 33032124
- [Background] Soffin EM, Beckman JD, Tseng A, Zhong H, Huang RC, Urban M, Guheen CR, Kim HJ, Cammisa FP, Nejim JA, Schwab FJ, Armendi IF, Memtsoudis SG. Enhanced Recovery after Lumbar Spine Fusion: A Randomized Controlled Trial to Assess the Quality of Patient Recovery. Anesthesiology. 2020 Aug;133(2):350-363. doi: 10.1097/ALN.0000000000003346. PMID 32433277
- [Background] Susano MJ, Scheetz SD, Grasfield RH, Cheung D, Xu X, Kang JD, Smith TR, Lu Y, Groff MW, Chi JH, Crosby G, Culley DJ. Retrospective Analysis of Perioperative Variables Associated With Postoperative Delirium and Other Adverse Outcomes in Older Patients After Spine Surgery. J Neurosurg Anesthesiol. 2019 Oct;31(4):385-391. doi: 10.1097/ANA.0000000000000566. PMID 30531557
- [Background] Susano MJ, Grasfield RH, Friese M, Rosner B, Crosby G, Bader AM, Kang JD, Smith TR, Lu Y, Groff MW, Chi JH, Grodstein F, Culley DJ. Brief Preoperative Screening for Frailty and Cognitive Impairment Predicts Delirium after Spine Surgery. Anesthesiology. 2020 Dec 1;133(6):1184-1191. doi: 10.1097/ALN.0000000000003523. PMID 32898243
- [Background] Waelkens P, Alsabbagh E, Sauter A, Joshi GP, Beloeil H; PROSPECT Working group * * of the European Society of Regional Anaesthesia and Pain therapy (ESRA). Pain management after complex spine surgery: A systematic review and procedure-specific postoperative pain management recommendations. Eur J Anaesthesiol. 2021 Sep 1;38(9):985-994. doi: 10.1097/EJA.0000000000001448. PMID 34397527